CLINICAL TRIAL: NCT00507845
Title: Use of Ramipril and Felodipine Combination Therapy in Hypertension: An Effectiveness Study With Local Patients in Argentina
Acronym: RAFEHELP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAMIP_L_01961
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Drug: Ramipril-Felodipine — Ramipril + felodipine 2.5/2.5mg per tablet. One tablet to be taken Od for 8 weeks (this dose could be increased at week 2 to 4 to 5 mg daily because of uncontrolled hypertension).
  Other Names: Triacor

SUMMARY:
Primary:

* To assess effectiveness of Ramipril-Felodipine in hypertensive Argentinean patients

Secondary:

* To assess tolerability of Ramipril-Felodipine in hypertensive Argentinean patients.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* Patients who couldn´t control their hypertension after 6 weeks of treatment with monotherapy (calcium blockers, beta blockers, diuretics, ACE inhibitors, AT2 blockers)(uncontrolled hypertension).

Exclusion Criteria:

* Already on fixed-dose combination treatment for hypertension
* Contraindication to angiotensin converting enzyme (ACE) inhibitors or CCB therapy
* Known hypersensitivity to felodipine (or other dihydropyridines), ramipril, other ACE or any of the excipients of ramipril felodipine.
* History of angioedema
* Unstable haemodynamic conditions: cardiovascular shock, untreated heart failure, acute myocardial infarction, unstable angina pectoris, stroke.
* Patients with AV block II or III
* Severely impaired hepatic function.
* Pre-existing bilateral renal artery stenosis or stenosis of the artery to a solitary kidney
* Pregnant and lactating mothers
* Patients on dialysis or haemofiltration.
* Patients with creatinine clearance < 20ml/min
* Use of potassium sparing diuretics
* Severe hypertension (SBP ≥ 180 mmhg or DBP ≥ 110 mmhg)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Mean changes in Systolic Blood Pressure (SBP) | from baseline to Week 8

SECONDARY OUTCOMES:
Mean changes in Diastolic Blood Pressure (DBP) | from baseline to Week 8
Percentage of responders with regard to DBP and SBP | comparison to baseline
Adverse events | After treatment and at each follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Cristian von Schulz Hausmann, MD, Study Director — Sanofi
Locations (1):
- Sanofi-aventis administrative office, Buenos Aires, Argentina